CLINICAL TRIAL: NCT05717777
Title: Treatment of Exertional Heatstroke witH icE wAter Soaked Towels
Acronym: THE HEAT
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Amber Hoek, Principal Investigator, Emergency Physician, MD, PhD, Erasmus Medical Center
Other Study IDs: 9805
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Heat Stroke Exertional; Heat Illness; Heat Exhaustion
MeSH Terms: conditions — Heat Stress Disorders; Heat Exhaustion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: There is no intervention, only observational study — There is no intervention, only observational study

SUMMARY:
Exertional heat stroke (EHS) is the most serious form of heat-illness that can occur during sports and exercise. If not recognized and treated immediately mortality rate of EHS is high. Early recognition and initiation of cooling are paramount. If temperature is reduced to < 40°C within 30 minutes of symptom onset, most patients recover completely. There are several strategies for cooling in EHS, including cooling with rotating in ice water soaked towels which cover the body of a patient.

The aim of this research is to investigate the effectiveness and safety of treatment of EHS with ice water soaked towels to lower body temperature.

DETAILED DESCRIPTION:
Rationale: Exertional heat stroke (EHS) is the most serious form of heat-illness that can occur during sports and exercise. If not recognized and treated immediately mortality rate of EHS is high. Early recognition and initiation of cooling are paramount. If temperature is reduced to < 40°C within 30 minutes of symptom onset, most patients recover without sequelae. Exertional heat exhaustion (EHE) is a precursor of EHS, and might develop in EHS if exercise is not terminated. There are several strategies for cooling in EHS, including cooling with rotating in ice water soaked towels which cover the body of a patient.

Objective: The aim of this research is to investigate the effectiveness and safety of treatment of EHS with ice water soaked towels to lower body temperature. Secondary objectives include cooling rate of ice water soaked towels, morbidity of EHS and HE, productivity loss related to EHS and EHE and the development of posttraumatic stress symptoms and PTSD after treatment for EHS and EHE.

Study design: We will conduct a prospective longitudinal observational study. Patients will be monitored and treated according the national guideline in the medical facility. A follow-up survey will be performed after two weeks and two months.

Study population: All participants of 18 years and older who received medical care for EHS or EHE at the City Pier City race on March 12th 2023 and Rotterdam Marathon on April 16th 2023.

Main study parameters/endpoints: Primary outcome will be the cooling rate of treatment with rotating in ice water soaked towels. Secondary outcomes will be percentage of patients with EHS that were cooled to a temperature lower than 40°C within 30 minutes after entering a medical facility (or collapse).

Hypothesis: Cooling with rotating in ice water soaked towels is an effective method for cooling patients with EHS by reducing the body temperature < 40°C within 30 minutes after symptoms.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There will be no risk from participating in the study and the burden will be low. The questionnaire will take approximately 20-30 minutes at two weeks and two months and 15 minutes at six months.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* ≥18 years
* Receive medical care at in the medical facility the City Pier City and Marathon Rotterdam 2023
* Tympanic temperature >38.0°C

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

• Language barrier (not proficient in Dutch or English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult runners who received medical care for EHS of EHE in the medical facility at the running events organized by Golazo Sports® at the City Pier City and Marathon Rotterdam 2023.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
cooling rate | during treatment in medical facility up to 2 hours after entering the facility
  cooling rate of treatment with rotating in ice water soaked towels

SECONDARY OUTCOMES:
percentage cooled to a temperature <40°C within 30 minutes | 30 minutes after entering medical facility
  be percentage of patients with EHS that were cooled to a temperature lower than 40°C within 30 minutes after entering a medical facility (or collapse).
Morbidity of EHS/EHE | 2 weeks and 2 months after EHS/EHE
  Morbidity of EHS and HE, clinical disease measured by questionnaires
productivity loss (abscens of work) related to EHS and EHE | 2 months after EHS/EHE
  Productivity loss measured by abscens of work questionnaire
Posttraumatic stress symptoms after EHS and EHE | 6 months after EHS/EHE
  Posttraumatic stress symptoms and PTSD after treatment for EHS and EHE by PCL-5 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No